CLINICAL TRIAL: NCT02361957
Title: The Effect of the Multispecies Probiotic Ecologic 825 Versus Placebo in Ulcerative Colitis Patients
Acronym: CUPIDO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: We recruited 25 of the 40 participants from intended study population. Recruitment in new populations requires an METC amendment.
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NL46674.081.13
Record Dates: First submitted 2015-01-15; First posted 2015-02-12 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator): Multispecies probiotic product Ecologic 825, 2x10-9 colony forming units per gram, 6 grams per day.
  Interventions: Dietary Supplement: Ecologic 825
- Placebo (Placebo Comparator): Similar in appearance as the probiotics, but not containing any bacteria.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ecologic 825 — Multispecies probiotic product, 2.5 x10E9 colony forming units per gram, 6 grams a day
  Other Names: PRO.IB
  Arms: Probiotics
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: The underlying etiology in inflammatory bowel diseases such as Ulcerative Colitis is not yet fully understood. Studies suggest a relation between higher intestinal permeability and aberrant changes of the epithelium. Dysbiosis of the intestinal microbiota might be the cause. Probiotics may restore the balance of the intestinal microbiota. In theory this could improve intestinal permeability and therefore reduce disease activity and maintain remission in patients with Ulcerative Colitis.

OBJECTIVE: To investigate whether a specifically designed multispecies probiotic mixture (ecologic 825®), as adjuvant therapy, can contribute to an improvement of intestinal permeability, microbiota composition, disease activity and inflammatory markers in ulcerative colitis.

STUDY DESIGN: 12-wk placebo-controlled randomized double-blind intervention with 2 parallel arms.

STUDY POPULATION: Adults diagnosed with left sided Ulcerative Colitis or Pancolitis in remission or mild stage of the disease. For inclusion of the patients the Patient Simple Clinical Colitis Activity Index (P-SCCAI) will be used.

INTERVENTION: Patients will receive either two daily dosages of 3 g of Ecologic® 825 or two daily doses of 3 g of the placebo, containing only the carrier material (both produced by Winclove Probiotics).

MAIN STUDY PARAMETERS/ENDPOINTS: Main study parameter is intestinal permeability measured by several techniques: the lactulose/mannitol absorption test (L/M test), LPS levels in blood serum and faecal zonulin. Secondary, inflammation will be measured from faecal calprotectin and blood c-reactive protein (CRP) levels. Furthermore samples will be stored to measure cytokine concentrations in serum and to analyse the microbial composition of the faecal samples using the HITchip. For the disease related quality of life the irritable bowel disease questionnaire (IBD-Q) and SF-36 will be used. All parameters will be measured at three time points; t=0, t=6 and t=12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Ulcerative Colitis (left sided UC or pancolitis)
* Age 18-65 (because microbiota change at older age)
* Stable disease activity (clinical remission with CRP levels <10mg/L and calprotectin <100 ug/g) as measured at baseline
* Mild disease activity (P-SCCAI <5)
* Mesalazine medication as only medication for UC with a maximum intake of 2.4 g/day

Exclusion Criteria:

* History of intestinal surgery that might interfere with the outcome of the study
* Diabetes Mellitus (medication dependent)
* Current use of antibiotics
* Current use of corticosteroids (30 days prior to the first baseline measurement).
* Treatment with other medication besides mesalazine (NSAIDs, topical or systemic steroids, immunosuppressive drugs or aspirin) one week prior the first baseline measurement.
* Use of other pre- and probiotics and not willing to stop these 2 weeks before the intervention period
* Hypersensitivity or allergy to milk protein, soy protein and gluten
* Alcohol abuse (male more than 14 servings a week, female more than 7 servings a week)
* Female patients: currently pregnant or breast-feeding or intending to become pregnant during the study
* Patients foreseen to need GI surgery during the study period
* Patients with a history of cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Intestinal permeability measured by the Lactulose Mannitol test (L/M test) | 12 weeks
  Measured by the Lactulose Mannitol ratio in urine (L/M test)

SECONDARY OUTCOMES:
blood CRP levels | 6 and 12 weeks
  inflammatory marker
fecal calprotectin levels | 6 and 12 weeks
  marker of intestinal inflammation
Quality of life (measured by IBD-Q and SF36) | 6 and 12 weeks
  Disease related quality of life will be measured by IBD-Q and SF36
Intestinal permeability measured by the Lactulose Mannitol test (L/M test) | 6 weeks
  Measured by the Lactulose Mannitol ratio in urine (L/M test)
Lipopolysaccharides levels in blood | 6 and 12 weeks
  A marker for intestinal permeability and inflammation
Intestinal permeability measured by faecal zonulin levels | 6 and 12 weeks
  Measured by faecal zonulin levels
microbiota composition | 6 and 12 weeks
  measured by human intestinal tract (HIT-chip) microarray
interferon gamma levels | 6 and 12 weeks
  measured in plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Nicole De Roos, PhD, Principal Investigator — Wageningen UR
Locations (1):
- Gelderse Vallei Hospital, Ede, Netherlands